CLINICAL TRIAL: NCT02046577
Title: A Randomized, Double-blind, Controlled Trial of Vitamin D for the Prevention of Acute Respiratory Infections in Children Aged 18 to 36 Months in Santiago, Coyhaique and Punta Arenas, Chile
Brief Title: Study of Vitamin D for the Prevention of Acute Respiratory Infections in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: National Fund for Research and Development in Health, Chile (Other); Laboratorio Pasteur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-116; Fonis SA13I20173 (Other Grant/Funding Number: Fondo Nacional de Investigación y Desarrollo en Salud)
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Acute Respiratory Tract Infections
Keywords: Acute respiratory tract infections; vitamin D; cholecalciferol; children; bronchiolitis; pneumonia; prevention
MeSH Terms: conditions — Bronchiolitis; Pneumonia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5600 IU Vitamin D3 (Experimental): Oral 5600 IU Vitamin D3 in liquid weekly during 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Oral 11200 IU Vitamin D3 weekly (Experimental): Oral 11200 IU Vitamin D3 in liquid weekly during 6 months
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Oral placebo in liquid weekly during 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Cholecalciferol administration
  Other Names: Cholecalciferol
  Arms: 5600 IU Vitamin D3; Oral 11200 IU Vitamin D3 weekly
Dietary Supplement: Placebo — Placebo liquid
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine whether weekly oral vitamin D supplementation is effective to prevent acute respiratory tract infections in children. The hypothesis of the study is that vitamin D supplementation reduces the incidence and severity of acute respiratory tract infections in children.

DETAILED DESCRIPTION:
Acute respiratory tract infections (ARTIs) are associated with high levels of morbidity and socioeconomic impact, particularly affecting young children. Observational studies have shown an association between vitamin D (VD) deficiency and higher incidence and severity of respiratory infections. Chile has a high prevalence of VD deficiency, particularly in the southern regions of the country. The objective of this study is to evaluate the safety and efficacy of oral VD supplementation to decrease the incidence of ARTIs in 275 preschool children. A randomized, placebo-controlled, double-blind study will be performed in Santiago, Coyhaique and Punta Arenas. Children aged 18 to 36 months will be given weekly oral 5600 IU of vitamin D3 (VD3), 11200 IU of VD3, or placebo doses during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 18 to 36 months attending daycare in Santiago, Coyhaique or Punta Arenas.

Exclusion Criteria:

* History of chronic illness requiring immunosuppression
* History of metabolic bone disease
* Use of vitamin D supplementation greater than 400 IU daily, either by milk formula or vitamin supplements in the last 3 months.
* Use of fish oil supplements in the last 3 months.
* Immunodeficiency
* Planned trip to sunny climate during study period.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of acute respiratory tract infections | 6 months

SECONDARY OUTCOMES:
Adverse events | 6 months
Hospitalizations due to acute respiratory tract infections | 6 months
Serum cathelicidin levels | 6 months
  Baseline and after 6 months measurement of serum cathelicidin levels.
serum 25-hydroxyvitamin D levels | 6 months
  Baseline and after 6 months measurement of serum 25-hydroxyvitamin D levels.
Viral etiology of ARTIs | 6 months
  Specific virological etiology of ARTIs will be evaluated by polymerase chain reaction in children with febrile ARTIs and with medical diagnosis of bronchiolitis or pneumonia.
Bone metabolism parameters | 6 months
  Baseline and after 6 months measurement of serum parathormone (PTH), alkaline phosphatases, calcium, phosphorus, and urinary calcium/creatinine ratio.

CONTACTS AND LOCATIONS:
Overall Officials: María L Reyes, M.D., Principal Investigator — Pontificia Universidad Catolica de Chile; Cecilia Vizcaya, M.D., Study Director — Pontificia Universidad Catolica de Chile; Arturo Borzutzky, M.D., Study Director — Pontificia Universidad Catolica de Chile; Catalina Le Roy, M.D., Study Director — Pontificia Universidad Catolica de Chile; Carlos A. Camargo Jr., M.D. Dr.PH., Study Director — Massachusetts General Hospital, Harvard University; Karin Brikmann, M.D., Study Director — Hospital Regional de Punta Arenas; Flavia Chamorro, M.D., Study Director — Hospital de Coyhaique; Marco Reyes, M.D., Study Director — Hospital de Coyhaique; Carolina Loureiro, M.D., Study Director — Pontificia Universidad Catolica de Chile
Locations (3):
- Chile (3):
  - Hospital de Punta Arenas, Punta Arenas, Region of Magallanes
  - Hospital Las Higueras, Talcahuano, Región del Biobío
  - Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided